CLINICAL TRIAL: NCT03139825
Title: Connectivity and Social Cognition in Adolescent Girls With Borderline Personality Disorder, a Pilot Study
Acronym: EEG-NIRS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not accepted
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0026
Record Dates: First submitted 2017-04-28; First posted 2017-05-04 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Adolescent Behavior; Borderline Personality Disorder
MeSH Terms: conditions — Adolescent Behavior; Borderline Personality Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescent with suicidal behavior and personality disorder (Other)
  Interventions: Other: Exploring the feasibility of learning during cognitive tasks (EEG-NIRS)

INTERVENTIONS:
Other: Exploring the feasibility of learning during cognitive tasks (EEG-NIRS) — Exploring the feasibility of the study in its aspects of recruitment and tolerability of tasks and acquisition of electrical and hemodynamic data that can be used during cognitive tasks

SUMMARY:
The disruption of social cognition associated with borderline personality disorder (BPD), and more specifically categorization of facial emotions, remains largely under-studied, despite the high frequency of this pathology in the clinical population. The first results differ from the observations made in adults and this confirms the relevance of studying this theme specifically in adolescence. On the cognitive level, there is a disturbance of the detection and the categorization of the facial emotions in the TPL. The characteristics of this disturbance and its possible association with an attack on the connectivity of the brain remain unknown in adolescence. No functional imaging studies are published in adolescent TPL. This pilot bimodal functional imaging study EEG-NIRS aims to collect preliminary and feasibility data to support a response to upcoming PHRC competitions and eventually offer a science thesis opportunity.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents 14-17 years of age with suicidal behavior and a borderline personality disorder for whom consent is obtained from parental authority,
* Affiliation to Social Security

Exclusion Criteria:

* Intellectual disability, psychopathy, delusional or concomitant major depression

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2018-02-22 (Estimated); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Analysis by functional imaging study of the characteristics of disorders of personalities and its possible association with an attack on connectivity of the brain | 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France